CLINICAL TRIAL: NCT04979741
Title: Recovery After Intensive Care Study: a Single- Center Observational Study
Brief Title: Recovery After Intensive Care Study
Acronym: RAI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Professor, University of Genova
Other Study IDs: CER Liguria: 350/2019; Protocol approval (Other: Genova)
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Follow up; Outcome; Intensive Care Unit Syndrome
Keywords: intensive care unit; cognitive dysfunction; delirium
MeSH Terms: conditions — Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — Observational study, no intervention is required

SUMMARY:
Post-ICU long term sequelae- defined as "post intensive care syndrome" (PICS) manifest with a wide spectrum of psychological and cognitive impairments, affecting over two-thirds of ICU survivors and leading to increased rehospitalization, health care costs, impaired quality of life (QoL), inability to return to work and burden for families.

The prevalence of post-traumatic stress symptoms (PTSD), anxiety symptoms, and depression after ICU stay is high and has been demonstrated in up to 50% of post-ICU population.

Therefore, over the last years, an important effort has been made for the development of ICU aftercare and follow-up clinics with the aim to detect and to minimize post-ICU sequelae and improve outcomes. However, the utility of these follow-up programs and their effect on outcome has not been completely demonstrated.

DETAILED DESCRIPTION:
This is a single center, prospective observational study, which will be conducted at Policlinico San Martino Hospital, Genova, Italy. Patients admitted to the ICU from more than 72 hours will be consecutively included during a 2 years period.

The primary objective is to assess the incidence of post-discharge mortality in patients admitted in ICU at 12 months.

Secondary objectives include the evaluation at 3, 6 and 12 months of outcome of patients admitted in ICU assessing QoL, anxiety, depression, PTSD, physical ability, cognitive function, sleep disorder and return to previous life; Self- and observer reported cognitive disability at 6 and 12 months after ICU discharge; prognostic factors for poor outcome, and emotional and burden of care impact on the patient's caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* All patients acutely admitted in the ICU from >72 hours, for both medical and surgical pathologies.

Exclusion Criteria:

* Pregnancy;
* Refuse of consent to enrolment of patient or of the doctor required to give his approval.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU from more than 72 hours will be consecutively included during a 2 years period
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of post-discharge mortality in patients admitted in ICU. | 12 months
  using a neuropsychological evaluation

SECONDARY OUTCOMES:
Cognitive outcome assessed through the MoCA scale, Montreal Cognitive Assessment | 12 months
  This is a scale including different tests regarding language, attention, naming giving a score from 0 (maximal cognitive dysfunction) and 30 ( no deficit)
Cognitive outcome assessed through HADS scale (Hospital Anxiety and Depression Scale) | 12 months
  Questionnaire with score from 0 (no issues) to 21 (maximal abnormalities) exploring depression and anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available for reasonable request to the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Request to the PI